CLINICAL TRIAL: NCT06236334
Title: The Validation of a Proof-of-concept Study of People at Risk for Diabetes With Personalised Lifestyle Interventions and E-health to Change Lifestyle Behaviour and Reverse the Risk for Diabetes
Brief Title: ELFI Health (e-Health for Empowerment by Lifestyle, Food Advice and Interaction)
Acronym: ELFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Roche Diagnostics GmbH (Industry); World Data Exchange (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9885 (TNO); NL85760.028.23 (Registry Identifier: ToetsingOnline The Netherlands); P2341 (Other: Ethical Review Board Brabant, The Netherlands)
Record Dates: First submitted 2024-01-12; First posted 2024-02-01 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pre-diabetes
Keywords: lifestyle; e-health; behavior
MeSH Terms: conditions — Glucose Intolerance; Behavior

STUDY DESIGN:
Intervention Model Description: People at risk for diabetes will be selected. Screening at HbA1c level will be a selection criterion
Masking Description: All subjects will participate in a blended/hybrid intervention of live and online lifestyle support
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle intervention (Experimental): The intervention will be a twelve week lifestyle intervention (live and online)
  Interventions: Behavioral: ELFI lifestyle intervention

INTERVENTIONS:
Behavioral: ELFI lifestyle intervention — A (digital) lifestyle support intervention. Based on anthropometrics, food intake and lifestyle preferences, subjects will receive behavioral lifestyle support, especially with the focus on healthy food intake.

SUMMARY:
In the present study the investigators will examine whether people living with prediabetes benefit from an e-health lifestyle intervention of three months.

DETAILED DESCRIPTION:
In the Netherlands about 1,2 million people are living with type 2 diabetes. This number increases weekly by an average of 1000 people. Besides, an equal number of people are living in a condition of prediabetes. In this precondition of type 2 diabetes, prevention is still possible for people by changing their lifestyle. Ideally, for every individual a personalised lifestyle intervention, adapted to the individual situation, biology and preferences is advised. A personalised lifestyle intervention is effective in preventing and delaying progression to type 2 diabetes. In this study, it will be investigated whether it is feasible to perform a personalised lifestyle intervention in combination with an online e-health platform. The e-Health for Empowerment by Lifestyle, Food advice and Interaction (ELFI) Health lifestyle intervention aims to improve the lifestyle of people with prediabetes to prevent them from developing type 2 diabetes.

Therefore, the primary objective is to execute a feasibility study of the ELFI Health lifestyle intervention for three months in people with prediabetes in primary care (based on HbA1c). The secondary objectives are assessing the impact of the ELFI health lifestyle intervention after three months on objective outcome parameters, including lipid profile, body composition, waist and hip circumference, blood pressure, and nutritional intake, as well as evaluating the lifestyle intervention and the online e-health platform used by participants and medical professionals.

The study is a feasibility study, studying the ability of a personalised lifestyle intervention and e-health platform to change lifestyle behaviour and decrease the risk for the development of type 2 diabetes in people with prediabetes.

The participants are newly diagnosed adults with prediabetes, aged 18-70 years. Prediabetes is defined as people with disturbed glucose values based on HbA1c levels of 39 - 53 mmol/mol (= 5.7 - 7.0%).

The intervention in this study consists of a personalised lifestyle intervention for three months. After measurements of HbA1c, blood lipids, body composition, waist and hip circumferences, blood pressure, and after assessment of food intake, a personal goal is set and participants start following the personalised lifestyle intervention. This is partly a digital intervention and partly a physical intervention (blended care). The digital part is followed via an online e-health platform, which offers different information modules. The physical part consists of different measurements of the outcome parameters and community events, where participants are in contact with their general practitioner and peers. Besides, participants have three appointments during the intervention period with a dietician to discuss their personalised program.

The main study outcome is the feasibility of the ELFI Health lifestyle intervention for three months in people with prediabetes in primary care. Key question is whether the intervention is appreciated by the subjects and working sufficiently to motivate participants in maintaining a healthier lifestyle. The feasibility will be evaluated by examination of the HbA1c level and subsequent prediabetes risk.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed with screening questionnaire
2. HbA1c: 39 - 53 mmol/mol (= 5.7 - 7.0%)
3. Age between 18 - 70 years
4. Stable BMI of 25 - 35 kg/m2
5. Informed consent signed
6. Willing to comply with the study procedures during the study
7. Being able to become more physically active, as assessed by the screening questionnaire (P9885 F02; in Dutch).
8. Being digitally competent
9. Willing to accept the use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years

Exclusion Criteria:

1. Being diagnosed with diabetes type 1 or 2
2. Use of insulin, corticosteroids (systemic), or beta-blockers in past month
3. Use of oral diabetes medication in past year
4. (Having a history of a) medical condition that might significantly affect the study outcome as judged by the general practitioner and health and lifestyle questionnaire. This includes gastrointestinal dysfunction, diseases related to inflammation or allergy, or a psychiatric disorder
5. Being abroad or on vacation for longer than a week.
6. Alcohol consumption > 21 (women) - 28 (men) units/week
7. Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
8. Recent blood donation (<1 month prior to the start of the study)
9. Not willing to give up blood donation during the study
10. Not willing to accept information-transfer concerning participation in the study, or information regarding his health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.
11. Pregnant or lactating women
12. Involved in another Combined Lifestyle Intervention or weight loss program
13. On GLP-1 analogues to stimulate weight loss

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Diabetes risk based on HbA1c level (mmol/mol) | three months
  Change in HbA1c due to lifestyle intervention (in mmol/mol)

SECONDARY OUTCOMES:
Lipid profile (mmol/L) | three months
  change in lipid profile due to lifestyle intervention (mmol/L)
body weight (kg) | three months
  change in body weight (kg) due to lifestyle intervention
body fat % (%) | three months
  change in body fat % (%) due to lifestyle intervention
waist circumference (cm) | three months
  change in waist circumference (cm) due to lifestyle intervention
hip circumference (cm) | three months
  change in hip circumference (cm) due to lifestyle intervention
Habitual food intake (frequencies, number and grams) | three months
  Changes in habitual food intake (frequencies, number and grams)will be examined with q food intake questionnaire before, during and after the intervention intervention program

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Wopereis, PhD, Principal Investigator — TNO
Locations (1):
- TNO, Leiden, Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uusitupa M, Khan TA, Viguiliouk E, Kahleova H, Rivellese AA, Hermansen K, Pfeiffer A, Thanopoulou A, Salas-Salvado J, Schwab U, Sievenpiper JL. Prevention of Type 2 Diabetes by Lifestyle Changes: A Systematic Review and Meta-Analysis. Nutrients. 2019 Nov 1;11(11):2611. doi: 10.3390/nu11112611. PMID 31683759
- [Background] Galaviz KI, Weber MB, Suvada K BS, Gujral UP, Wei J, Merchant R, Dharanendra S, Haw JS, Narayan KMV, Ali MK. Interventions for Reversing Prediabetes: A Systematic Review and Meta-Analysis. Am J Prev Med. 2022 Apr;62(4):614-625. doi: 10.1016/j.amepre.2021.10.020. Epub 2022 Feb 10. PMID 35151523